CLINICAL TRIAL: NCT03525145
Title: Platelet Reactivity And Clinical ThrombotIC Events Study
Acronym: PRACTICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Prof., Shenyang Northern Hospital
Other Study IDs: PRACTICEV1.02
Record Dates: First submitted 2018-04-25; First posted 2018-05-15 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Acute Coronary Syndrome; Antiplatelet Therapy; Platelet Reactivity
Keywords: Platelet Reactivity; Thrombotic Events
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Platelet function testing has been considered for DAPT strategy adjustments to reduce the patient's risk of ischemia and bleeding. Although several previous RCT studies did not find any benefit in the detection of platelet function， the previous studies were mostly low-risk populations, and the P2Y12 receptor antagonists were simply clopidogrel, and the detection methods were relatively simple. Therefore, the need for platelet monitoring in high-risk ACS patients receiving new potent P2Y12 inhibitor ticagrelor, as well as the diagnostic threshold for different platelet function assays needs further study. In addition, due to the differences on the response to anti-platelet drugs between the East and the West, it is not appropriate to simply refer to the conclusion of the other party. However, as of now, there is no large sample randomized controlled study systematically focused on the applicability and status of platelet function tests in East Asian populations, especially Chinese populations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. There was a history of at least one acute coronary syndrome (ACS) attack within 14 days before enrollment, including unstable angina, non-ST elevation myocardial infarction, or ST-elevation myocardial infarction;
3. Being treated with aspirin and a P2Y12 inhibitor (clopidogrel or ticagrelor);
4. Plan to apply dual antiplatelet drugs (DAPT, aspirin + P2Y12 inhibitor) for at least 12 months;
5. Voluntary signature of informed consent

Exclusion Criteria:

1. In combination with other anti-platelet drugs, such as cilostazol;
2. Have received glycoprotein IIb/IIIa inhibitor within 72 hours before enrollment;
3. receving a P2Y12 inhibitor loading does less than 72h or maintenance (unloaded) less than 5d;
4. Plan to perform any coronary revascularization within 30 days;
5. The need for oral anticoagulants (warfarin, factor II or factor X inhibitors);
6. Predicted survival time <12 months for patients with known severe progressive disease (such as malignancy) or extreme depletion of the disease;
7. pregnant women or pregnant people;
8. Any situation that may interfere with the research process, such as dementia, delirium, alcoholism, etc.;
9. expected to undergo surgery within 1 year;
10. Patients participating in other ongoing clinical studies

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome undergoing antiplatelet therapy
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular thrombotic events | One Year
  Cardiovascular death, non-fatal myocardial infarction, stroke, or stent thrombosis

SECONDARY OUTCOMES:
Cardiovascular death | One Year
  Cardiovascular death
BARC(Bleeding Academic Research Consortium )2-5 Bleeding | One Year
  BARC2-5 Bleeding
MACCE(Major adverse cardiac and cerebral events) | One Year
  Cardiovascular death, non-fatal myocardial infarction, stroke, or ischemic-driven target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Study Director — Northern Hospital
Locations (1):
- Northern Hospital, Shenyang, Liaoning, China